CLINICAL TRIAL: NCT05392309
Title: Effects of Manual Ankle Rocking Training on Postural Control and Foot Function in Children With Down Syndrome
Brief Title: Manual Ankle Rocking Training on Postural Control and Foot Function in Children With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0704
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Down S Syndrome
Keywords: Down syndrome; Postural control; Postural stability; Balance
MeSH Terms: conditions — Down Syndrome | interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual ankle rocking training (Experimental): Group will receive manual ankle rocking training with lower limb exercise and core strengthening of trunk
  Interventions: Other: Manual ankle rocking training; Other: Conventional
- conventional (Active Comparator): Group will receive lower limb exercises and core strengthening of trunk. Sessions will be 4 days in a week
  Interventions: Other: Conventional

INTERVENTIONS:
Other: Manual ankle rocking training — Group will receive manual ankle rocking training with lower limb exercise and core strengthening of trunk
  Arms: Manual ankle rocking training
Other: Conventional — Group will receive lower limb exercises and core strengthening of trunk. Sessions will be 4 days in a week

SUMMARY:
Down syndrome occurs due to abnormal cell division of extra chromosome 21. It is a genetic disorder that causes postural un stability, leads to poor foot function and causes them difficulty that they can't fulfill their daily life activities and can't be independent. Strengthening exercise of lower limb and core strengthening of trunk muscle will provide postural stability and lower limb strengthening. Aim of this research is to determine the effects of manual Ankle rocking training on postural control and foot function in children with Down syndrome. Those who are diagnosed with down syndrome and are between age 8-15 and both of the genders are included in this research and those who have any surgical issue, visual impairment and musculoskeletal contractures are not included in the study we will use static standing balance test to check postural control and foot function index for Ankle rocking training from two group in which one will be given the baseline treatment of lower limb exercise and core strengthening with ankle rocking training and the other group without ankle rocking training and then the collected data will be analyzed by SPSS. 22

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed children with down syndrome
* Age 8 to 15
* Both gender (male and female)

Exclusion Criteria:

* Musculoskeletal contractures
* Visual or other sensory input impairment
* Any surgical procedure

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Changes in foot function index score | Baseline and 9th week
  A Foot Function Index (FFI) was developed in 1991 to measure the impact of foot pathology on function in terms of pain, disability and activity restriction. It is a self-administered index consisting of 23 items divided into 3 sub-scales. Both total and sub-scale scores are produced.
Static standing balance test | baseline and 9th week
  Static standing balance test for postural control and stability

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Afzal, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Rising Sun Institute For Special Children, Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balan V, Georgescu M. Postural control in Down syndrome subjects. European Proceedings of Social and Behavioural Sciences. 2019;11.
- [Background] Palomba A, Perez D, Tafuri D. THE EFFECTS OF PHYSICAL ACTIVITY ON BALANCE AND POSTURAL CONTROL IN PEOPLE WITH DOWN SYNDROME.
- [Background] Shields N, Lim P, Wollersheim D, Nikolopoulos N, Barrett J, Evans A, et al. Do foot posture, deformity, and footwear fit influence physical activity levels in children with Down syndrome? A prospective cohort study. Journal of Intellectual & Developmental Disability. 2017;42(4):332-8
- [Background] Wang HY, Long IM, Liu MF. Relationships between task-oriented postural control and motor ability in children and adolescents with Down syndrome. Res Dev Disabil. 2012 Nov-Dec;33(6):1792-8. doi: 10.1016/j.ridd.2012.05.002. Epub 2012 Jun 13. PMID 22699252
- [Background] Zago M, Duarte NAC, Grecco LAC, Condoluci C, Oliveira CS, Galli M. Gait and postural control patterns and rehabilitation in Down syndrome: a systematic review. J Phys Ther Sci. 2020 Apr;32(4):303-314. doi: 10.1589/jpts.32.303. Epub 2020 Apr 2. PMID 32273655
- [Background] Eltohamy AM, Mahran MA, Elassal MI, Kamel AH. Ankle Rocking Training and Functional Abilities in Children with Cerebral Palsy. The Egyptian Journal of Hospital Medicine. 2021;85(1):3301-5
- [Background] Chen HL, Yeh CF, Howe TH. Postural control during standing reach in children with Down syndrome. Res Dev Disabil. 2015 Mar;38:345-51. doi: 10.1016/j.ridd.2014.12.024. Epub 2015 Jan 13. PMID 25590172
- [Background] Brugnaro BH, Oliveira MFP, de Campos AC, Pavao SL, Rocha NACF. Postural control in Down syndrome and relationships with the dimensions of the International Classification of Functioning, Disability and Health - a systematic review. Disabil Rehabil. 2022 Jun;44(11):2207-2222. doi: 10.1080/09638288.2020.1830439. Epub 2020 Oct 13. PMID 33049152